CLINICAL TRIAL: NCT04558606
Title: Efficacy of Philips Sonicare Flexcare Platinum Toothbrush® Compared to Manual Brushing in Healthy Patients: a 1 Year Follow up
Acronym: SONIMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Magda Mensi, Principal investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SONIMAN
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2019-01

CONDITIONS: Gingivitis
Keywords: Oral Hygiene; Dental Care Instruction
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Monocetric, pragmatic, single blinded, randomized clinical trial, parallel design.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonic toothbrush (Experimental): * All patients receive full periodontal charting, a session of professional oral hygiene and OHI (oral hygiene instruction).
  * Each patient is instructed by the hygienist in the correct use of the sonic toothbrush
  Interventions: Device: Sonic Toothbrush
- Manual toothbrush (Active Comparator): * All patients receive full periodontal charting, a session of professional oral hygiene and OHI (oral hygiene instruction).
  * Each patient is instructed by the hygienist in the correct use of the manual toothbrush
  Interventions: Device: Manual Toothbrush

INTERVENTIONS:
Device: Sonic Toothbrush — Sonic Toothbrush (Philips Sonicare Flexcare Platinum Toothbrush®)
  Arms: Sonic toothbrush
Device: Manual Toothbrush — Manual brushing (Technique Pro - GUM® Sunstar Italiana SRL)
  Arms: Manual toothbrush

SUMMARY:
Professional oral hygiene has become a customary procedure in everyday dentistry. Both manual and sonic brushes are part of normal oral hygiene education practice. Compared with manual toothbrushes, ergonomic instruments, such as sonic toothbrushes, can be a more practical and less demanding mean to remove biofilm and plaque efficiently. Studies in literature investigate the efficacy of toothbrushes in plaque removal, but the investiagator's study would validate efficacy of toothbrushes post-causal therapy, towards lower plaque accumulation, and reduction in bleeding.

The objective of this study is to compare two methods (manual VS sonic) of tooth brushing in terms of impact on the gingival index and plaque index after one session of Full Mouth-Erythritol Powder Air Polishing Therapy (FM-EPAPT) in healthy patients.

The hypothesis of the present randomized controlled trial is that sonic tooth brushing accumulates less plaque (-10%) than manual tooth brushing.

To test this hypothesis, the patients, upon initial evaluation, will be divided in 2 study groups and, after a session of professional oral hygiene, will be instructed to use:

* CONTROL: manual toothbrush
* TEST: sonic toothbrush. Gingival index and plaque score will be evaluated at 2, 4, 6 weeks and 6 and 12 months.

DETAILED DESCRIPTION:
Everyone's goal to have a healthy mouth is the removal of biofilm, plaque and calculus from the dental surface everyday. Moreover routine recalls ensure a better oral health and greater protection against caries, gingivitis and periodontitis. Regular attendance to oral hygiene sessions plays an important role but has to be accompanied by the compliance with home oral care instructions. The patients should be adequately instructed to take care of their oral health.

TRIAL DESIGN: Monocetric, pragmatic, single blinded, randomized clinical trial (RCT) of parallel design.The trial will have one-year duration.

STUDY POPULATION: Healthy subject affected by gingivitis are included in the study. Presence of gingivitis is defined as bleeding on probing (BOP) > 25%.

PRIMARY OUTCOME: Change in Plaque Index (PI): change in 10% less of the site in test group.

SECONDARY OUTCOME:

* Change in Gingival Index (GI): change in presence or absence of bleeding after gently run on the surface of the marginal gingiva.
* Change in Recession (REC): change in gingival reduction.
* Change in Clinical Attachment Level (CAL): change in clinical attachment level.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by gingivitis is defined as bleeding on probing (BOP) > 25%.
* Healthy young patients (18-40 years)
* Patients with almost 5 teeth per quadrant
* Patients smoking less than 10 cigarettes a day

Exclusion Criteria:

* Presence of periodontitis (pocket depth - PPD > 4 mm)
* Patient with BOP and/or plaque index < 25%
* Patient with any systemic disease
* Orthodontic or prosthesis patient
* Patient with split
* Impossibility to come to the recall appointments
* Not willing to follow the agreed protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Change in Plaque Index (PI) | Baseline, 2, 4, 6 weeks and 6, 12 months
  Change in percentage of site with plaque. Baseline values will be compared to the values recorded in the follow-up visits. Change in 10% of the site in test group. 10% site modification in favor of the test group.

SECONDARY OUTCOMES:
Change in Gingival Index (GI) | Baseline, 2, 4, 6 weeks and 6, 12 months
  Change in percentage of site with bleeding after gently run on the surface of the marginal gingiva. Baseline values will be compared to the values recorded in the follow-up visits.
Change in REC (Clinical Gingival Recession) | Baseline 6, 12 months
  Change in mean of REC value for each patient should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.
Change in CAL (Clinical Attachment Level) | Baseline 6, 12 months
  Change in mean of CAL value for each patient should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Mensi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Magda Mensi, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04558606/Prot_000.pdf